CLINICAL TRIAL: NCT06027164
Title: Kosmos Trio and Ejection Fraction Pivotal Study
Status: Completed | Type: Observational
Sponsor: EchoNous Inc. (Industry)
Collaborators: University of California, San Francisco (Other); Revival Research Institute LLC (Unknown); Centaur Labs (Unknown)
Responsible Party: Sponsor
Other Study IDs: ECHO-004
Record Dates: First submitted 2023-07-27; First posted 2023-09-07 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Study Subjects: Ultrasound scans conducted by novice users and experts on this cohort.
  Interventions: Device: Portable Ultrasound System

INTERVENTIONS:
Device: Portable Ultrasound System — EchoNous KOSMOS

SUMMARY:
This is a single-group, observational study which will involve obtaining two echo scans of recruited patients. All recruited patients will undergo echo scans by both novice users (nurses) and experts (echo sonographers). Image quality between novices and experts as well as the ability to calculate LVEF from novice and expert scans and the quality of the LVEF calculated via KOSMOS-EF compared to LVEF calculations by expert cardiologists will occur in post-hoc Echo image analysis

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-89 years of age
* Have capacity to provide written consent either themselves or via healthcare proxy as determined by subjects' clinical care teams
* Have an anticipated timeline in the EDOU long enough to allow for completion of study procedures without causing delay to subjects' usual clinical care

Exclusion Criteria:

* Heart rate > 110 beats per minute at the time of recruitment
* Pregnant women
* Prior chest surgery
* Chest wall deformities or injuries (i.e. wounds, infections, etc)
* Limited mobility precluding them from turning in bed independently
* Speak a primary language other than English or Spanish
* Vulnerable populations including: patients being evaluated for psychiatric crises, incarcerated individuals
* Unwilling or unable to consent to study procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Emergency Department Observation Unit (EDOU) will be eligible for enrollment. Patients admitted to the EDOU often spend a prolonged amount of time in the EDOU (often > 24 hours) awaiting further testing, therapies, or specialist consultations, thus recruiting from this pool of patients is most likely to allow for completion of study procedures without impacting the course of their clinical care
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Assessment of Global Left Ventricular Function | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  A panel of cardiologists will access and determine via a majority vote if a study exam acquired by a nurses is of sufficient image quality to make a qualitative visual assessment of the Global Left Ventricular Function.
Assessment of Left Ventricular Size | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  A panel of cardiologists will access and determine via a majority vote if a study exam acquired by a nurse is of sufficient image quality to make a qualitative visual assessment of the Left Ventricular Size.
Assessment of Non-Trivial Pericardial Effusion | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  A panel of cardiologists will access and determine via a majority vote if a study exam acquired by a nurse is of sufficient image quality to make a qualitative visual assessment of Non-Trivial Pericardial Effusion.
Assessment of Right Ventricular Size | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  A panel of cardiologists will access and determine via a majority vote if a study exam acquired by a nurse is of sufficient image quality to make a qualitative visual assessment of Right Ventricle Size.

SECONDARY OUTCOMES:
Assessment of Automatic Structure Labelling | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  A panel of cardiologists will access and determine via a majority vote if the frame-level false discovery rate (FDR) of automated cardiac structure labeling as determined by expert cardiologists for scans acquired by cardiac sonographers.
Manual vs. KOSMOS-EF for Sonographer Scans | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  Measurements are computed for A4C and A2C scans acquired by sonographers . We will compare KOSMOS-EF LVEF calculation to LVEF calculated by a panel of cardiologists via a majority vote.
Assessment of Left Atrial Size | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  A panel of cardiologists will access and determine via a majority vote if a study exam acquired by a nurse is of sufficient image quality to make a qualitative visual assessment of Left Atrial Size.

CONTACTS AND LOCATIONS:
Locations (1):
- Revival Research Institute LLC, Dearborn, Michigan, United States